CLINICAL TRIAL: NCT04323826
Title: Effect of the Type and Emulsification of Dietary Fat on the Bioavailability of Fat-soluble Nutrients in Human
Brief Title: Effect of the Type and Emulsification of Dietary Fat on the Carotenoids Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant professor, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: S10
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Carotenoids
Keywords: Carotenoids absorption; blood triglycerides; postprandial lipid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- salads with olive oil-water mixture (Experimental): Vegetable salads (100g tomatoes, 62g carrots, 70g spinach, 25g lettuce and 5g wolfberry) with 56g olive oil-water mixture will be provided to consume.
  Interventions: Other: olive oil-water mixture
- salads with olive oil-water emulsion (Experimental): Vegetable salads (100g tomatoes, 62g carrots, 70g spinach, 25g lettuce and 5g wolfberry) with 56g olive oil-water emulsion (4% whey protein isolate as emulsifier) will be provided to consume.
  Interventions: Other: olive oil-water emulsion
- salads with coconut oil-water emulsion (Experimental): Vegetable salads (100g tomatoes, 62g carrots, 70g spinach, 25g lettuce and 5g wolfberry) with 56g coconut oil-water emulsion (4% whey protein isolate as emulsifier) will be provided to consume.
  Interventions: Other: coconut oil-water emulsion
- salads with coconut oil-water mixture (Experimental): Vegetable salads (100g tomatoes, 62g carrots, 70g spinach, 25g lettuce and 5g wolfberry) with 56g coconut oil-water mixture will be provided to consume.
  Interventions: Other: coconut oil-water mixture

INTERVENTIONS:
Other: olive oil-water mixture — 50% olive oil in water, processed with high shear mixer at 8000 rpm power without adding emulsifier, well shaked before consumption.
  Arms: salads with olive oil-water mixture
Other: olive oil-water emulsion — 50% olive oil in water (4% whey protein isolate), stirred for 5 mins using a high shear mixer at 8000 rpm power and was further processed with high pressure homogenizer at 100 MPa.
  Arms: salads with olive oil-water emulsion
Other: coconut oil-water mixture — 50% coconut oil in water, processed with high shear mixer at 8000 rpm power without adding emulsifier, well shaked before consumption.
  Arms: salads with coconut oil-water mixture
Other: coconut oil-water emulsion — 50% coconut oil in water (4% whey protein isolate), stirred for 5 mins using a high shear mixer at 8000 rpm power and was further processed with high pressure homogenizer at 100 MPa.
  Arms: salads with coconut oil-water emulsion

SUMMARY:
This study is designed to assess the effects of 1) the emulsification 2) the type of dietary fat on carotenoid (CAT) absorption employing an in-vitro digestion system (Proof of Concept) and well-designed randomized controlled trial.

DETAILED DESCRIPTION:
In all, twenty-five healthy men and women (aged =19 and =45 y, approximately half men and half women, with the expectation that = 20 subjects will complete the study (= 20 % dropout rate)) will be recruited and each subject will participate in 4 trials (randomized and crossover). Anthropometric measurements, including height, weight, waist circumference, blood pressure as well as skin scan carotenoids status will be measured on the screening day as subject baseline information. Prior to each trial, subjects are required a compliance test (CT) visit. On that day, fasting blood will be drawn to analysis the CAT concentration and compare the analyzed CAT concentration to those of testing day baseline to assess the compliance of the washout diet period. Skin CAT scan status will also be conducted. After the CT day, subjects will undergo a 7-day washout period and follow low-CAT diet to reduce circulating, endogenous levels of CAT and minimize the contribution of CAT in the plasma. During the first 5 days, subjects will consume a low-CAT diet (CAT<750µg), and during the 6-7days, subjects will consume an even low-CAT diet (CAT<500µg). The low-CAT diet menu sheet will be provided and dietary instruction to achieve the low CAT diet will be given. Compliance with the low CAT diet will be promoted by daily menu check-off lists and in-person contact on visit day.Subject will be randomly assigned to consume a carefully portioned mix-vegetable salad (including tomatoes, shredded carrots, spinach, lettuce, and Chinese wolfberry) with 4 different oil-water combinations on the 4 meal testing (MT) day. The 4 different oil-water combinations are as follows:1) Olive oil-water mixture (non-emulsified, rich in unsaturated fat);2) Olive oil-water emulsification (rich in unsaturated fat);3) Coconut oil-water mixture (non-emulsified, rich in saturated fat);4) Coconut oil-water emulsification (emulsified, rich in unsaturated fat).On every MT day, fasting blood will be collected for analyzing the CAT levels every 60 minutes for 10 hours and CAT concentration, triglycerides will be analyzed from the collected blood samples. Appetite VAS questionnaire will be conducted every half hour in the first two hours after consuming test meal and hourly conducted till the 5th hour when lunch ( low-CAT (< 2000 µg), low-fat (<2 g)) provided. After consuming the lunch, Appetite VAS questionnaire will be conducted every half hour in the first two hours and hourly till the 10th hour. Thus, the timepoint for appetite VAS measurement will be at 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 9, 10 hour.There are no incidental findings in the current research as we will only collect subject's biological sample (blood) for testing the carotenoids level and blood triglycerides level which are the aim of this study. The rest measurements, including blood pressure, weight, height and waist circumference, they are the baseline information we collect for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give an informed consent
2. Age 19 to 45 years
3. Willing to follow the study procedures

Exclusion Criteria:

1. Significant weight change > 3 kg in the past 3 months;
2. Exercising vigorously over the past 3 months (*Defined as having > 6 metabolic equivalents of exercise daily; approximately 20 mins of moderate intensity exercise (e.g. slow jogging);
3. Intestinal disorders including lipid malabsorption;
4. Diabetes or prediabetes (fasting blood glucose > 100 mg/dL);
5. Smoking;
6. Drinking more than 2 alcoholic drinks per day;
7. Taking lipid-lowering medications or dietary supplements affecting plasma lipid-lipoprotein concentration.
8. Menopausal women, those using hormone based contraceptives, those having abnormal menstrual cycles, and those who are pregnant, lactating or planning to become pregnant.
9. Following any restricted diet (e.g. vegetarian)
10. Taking dietary supplements which may impact the outcome of interests (e.g. carotenoids supp.)
11. Insufficient venous access to allow the blood collection

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Blood carotenoids concentrations | Up to 6 months
  Five main carotenoids compounds, lutein, zeaxanthin, α-carotene, β-carotene and lycopene concentrations will be determined in blood via HPLC.
Blood triglycerides concentrations | Up to 6 months
  Plasma triglyceride concentration will be determined by using a Cobas c311 chemistry analyzer (Roche Diagnostics, Asia Pacific).

SECONDARY OUTCOMES:
Skin carotenoid status | Up to 4 months
  Measured using resonance Raman spectroscopy.
Height | Baseline data, up to 4 weeks
  Height (cm)
Weight | Baseline data, up to 4 weeks
  Weight (kg)
Waist circumference | Baseline data, up to 4 weeks
  waist circumference (cm)
Diet | Up to 6 months
  Dietary analysis via 3-day food record

CONTACTS AND LOCATIONS:
Overall Officials: KIM Jung EUN, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - Department of Food Science and Technology; National University of Singapore, Singapore
  - Investigational Medical Unit (IMU), Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JE, Gordon SL, Ferruzzi MG, Campbell WW. Effects of egg consumption on carotenoid absorption from co-consumed, raw vegetables. Am J Clin Nutr. 2015 Jul;102(1):75-83. doi: 10.3945/ajcn.115.111062. Epub 2015 May 27. PMID 26016861
- [Derived] Yao Y, Yang Z, Yin B, Goh HM, Toh DWK, Kim JE. Effects of dietary fat type and emulsification on carotenoid absorption: a randomized crossover trial. Am J Clin Nutr. 2023 May;117(5):1017-1025. doi: 10.1016/j.ajcnut.2023.03.011. Epub 2023 Mar 13. PMID 36921903